CLINICAL TRIAL: NCT01122225
Title: Neutrophile Gelatinase Associated Lipocalin Evaluation in Septic Acute Kidney Injury
Acronym: NESAKI
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Université Victor Segalen Bordeaux 2 (Other)
Collaborators: Inverness Medical Innovations (Industry)
Responsible Party: Fabrice CAMOU, MD, University Hospital of Bordeaux
Other Study IDs: NESAKI08-267
Record Dates: First submitted 2010-05-10; First posted 2010-05-13 (Estimated); Last update posted 2010-05-31 (Estimated); Status verified 2010-04

CONDITIONS: Acute Kidney Failure
Keywords: septic shock; medical intensive care
MeSH Terms: conditions — Acute Kidney Injury; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood Sample (350 µl) at inclusion and then 24 and 48 hours after
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Septic shock

SUMMARY:
Acute kidney injury (AKI) is a major organ failure in septic shock. Current medical tests (serum creatinine and urea) cannot identify AKI until approximately 48 hours after it occurs. Neutrophil gelatinase-associated lipocalin (NGAL) may be able to predict ischemic AKI more effectively and faster than serum creatinine and urea levels.

The purpose of this study is to take a blood sample from patients at admission and then at 24 and 48 hours after to test their plasma for NGAL and compare the NGAL levels to their creatinine and urea levels. The investigators hypothesize that NGAL is an earlier marker to classify the kidney failure as acute tubular necrosis or pre-renal azotemia than creatinine and urea.

DETAILED DESCRIPTION:
Primary Outcome Measures:

To correlate elevated serum NGAL with the diagnosis of intrinsic acute kidney injury in septic shock

Secondary Outcome Measures :

To compare serum NGAL with serum creatinine, serum urea and urine output in septic AKI Death within the intensive care unit Death from all causes at 28 days after inclusion

ELIGIBILITY:
Inclusion Criteria:

* Patients showing signs of infection and hypotension requiring the use of epinephrine despite of an appropriate fluid challenge.
* 18 years of age or older

Exclusion Criteria:

* Age under 18 years
* Prisoners or other institutionalized or vulnerable individuals
* Participation in an interventional clinical study within the previous 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients of a medical intensive care presenting with a septic shock
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-07; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice Camou, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Reanimation medicale, Hopital Saint-Andre, Bordeaux University Hospital, Bordeaux, Aquitaine, France